CLINICAL TRIAL: NCT06199128
Title: Evaluation of the Efficacy and Safety of the Local Treatment of Carboxymethyl Beta-glucan and Polycarbophil in Patients With Normal Cytology/ASCUS/LSIL (CIN1) With HPV+ PCR Determination
Brief Title: Efficacy and Safety of Carboxymethyl Beta-glucan and Policarbophil in HPV Positive Patients
Acronym: Fix
Status: Completed | Type: Observational
Sponsor: Uriach Consumer Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: The Fix Study V.2 12/Jul/2022
Record Dates: First submitted 2023-12-18; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Human Papillomavirus Infection
Keywords: HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CONTROL GROUP: For the duration of the study, standard clinical practice will be followed wait and see strategy, without administering carboxymethyl-b-glucan treatment.
- TREATMENT GROUP: For a period of three months, patients will be administered once daily treatment with Carboxymethyl β-glucan and Polycarbophil
  Interventions: Dietary Supplement: carboxymethyl β-glucan

INTERVENTIONS:
Dietary Supplement: carboxymethyl β-glucan — It is a vaginal spray gel designed for the prevention and treatment of cervical lesions caused by HPV. This is achieved by controlling the physiological conditions of the transformation zone of the cervico-vaginal mucosa. The composition of the gel, which includes polycarbophil and carboxymethyl-beta-glucan, effectively shields the cervico-vaginal mucosa from the damaging effects of external agents due to its bioadhesive capacity. Additionally, it contributes to the re-epithelialization and regression of cervical lesions
  Groups: TREATMENT GROUP

SUMMARY:
Prospective, Controlled, Multicentre, Real Clinical Practice Study. Effectiveness of Carboxymethyl β-Glucan treatment in high-risk HPV+ patients

DETAILED DESCRIPTION:
To evaluate the effectiveness of local treatment with carboxymethyl-b-glucan and polycarbophil on the clearance time of human papillomavirus (HPV), as well as on the normalisation of cytological alterations identified at study inclusion.

ELIGIBILITY:
TREATMENT GROUP

INCLUSION:

* Women aged between 25 and 65 years (inclusive).
* Histological cervical cytology results reported as ASCUS, LSIL/CIN1, with a positive cervical PCR determination for high-risk HPV (genotypes 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68).
* Patients currently undergoing treatment with the combination of carboxymethyl B-glucan and polycarboxyl (for at least 15 days prior to study initiation)
* Capable of reading and comprehending the patient information sheet and the informed consent form.
* Willing to participate in the study and sign the informed consent form.

EXCLUSION:

* Cervical cytology indicating suspected invasive cervical cancer.
* Ongoing or recent pregnancy terminated within six weeks of the study commencement.
* Clinically significant immunodeficiency-linked pathology.
* Active or terminated immunosuppressive treatment within six months of study entry. Specifically, in the case of corticosteroids, women will be excluded if they are currently or recently receiving corticosteroid treatment (defined as within two weeks prior to study entry) or if they have undergone two or more cycles of corticosteroids at doses equal to or greater than 20 mg/day of Prednisone (or equivalent) orally or parenterally for at least one week's duration in the year prior to study entry.
* Undiagnosed abnormal genital bleeding.
* Total hysterectomy.
* Documented history of cervical pathology caused by HPV.
* Contraindications to the use of the combination of Carboxymethyl B-glucan and polycarboxyl, or known allergies to any of its components.

CONTROL GROUP

INCLUSION:

* Women aged between 25 and 65 years (inclusive).
* Histological cervical cytology results reported as ASCUS, LSIL/CIN1, with a positive cervical PCR determination for high-risk HPV (genotypes 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68).
* Patients not currently undergoing treatment for HPV.
* Capable of reading and comprehending the patient information sheet and the informed consent form.
* Willing to participate in the study and sign the informed consent form.

EXCLUSION:

* Cervical cytology indicating suspected invasive cervical cancer.
* Ongoing or recent pregnancy terminated within six weeks of the study commencement.
* Clinically significant immunodeficiency-linked pathology.
* Active or terminated immunosuppressive treatment within six months of study entry. Specifically, in the case of corticosteroids, women will be excluded if they are currently or recently receiving corticosteroid treatment (defined as within two weeks prior to study entry) or if they have undergone two or more cycles of corticosteroids at doses equal to or greater than 20 mg/day of Prednisone (or equivalent) orally or parenterally for at least one week's duration in the year prior to study entry.
* Undiagnosed abnormal genital bleeding.
* Total hysterectomy.
* Documented history of cervical pathology caused by HPV.
* Concurrent participation in a clinical study of an investigational drug that could interfere with the current study.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The data will be collected from patients who meet the selection criteria.
Sampling Method: Probability Sample
Enrollment: 533 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Evolution in the total or partial negativization of high-risk HPV infection in women with or without cytological alterations upon local treatment with carboxymethyl-β-glucan and polycarbophil. | 6 months
  Evaluation of the total or partial negativization of HPV by HPV PCR test with genotype

SECONDARY OUTCOMES:
Normalization rate of abnormal colposcopy | 6 Months
  Evaluation of abnormal or normal colposcopy
Change in the incidence of cytological alterations upon local treatment with carboxymethyl - β-glucan and polycarbophil during the follow-up time | 6 Months
  Change in the incidence of cytological alterations development measured by reflex cytology test (Normal Cytology; ASCUS; LSIL or HSIL cytology)
Determine the effect of local treatment with carboxymethyl - β-glucan and polycarbophil on the total negativization rate of HPV | 6 Months
  Evaluation of HPV total negativization rate by HPV PCR test with genotype

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Pingarrón Santofima, Doctor, Principal Investigator — Hospital Quirón San José
Locations (5):
- Spain (5):
  - Hospital CIMA, Barcelona, Barcelona
  - Hospital Quirón San José, Madrid
  - Hospital Universitario Infanta Leonor,, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Quirón Donostia, San Sebastián

REFERENCES:
- [Background] Stentella P, Biamonti A, Carraro C, Inghirami P, Mancino P, Pietrangeli D, Votano S, Lazzari P, DE Medici C. Efficacy of carboxymethyl beta-glucan in cervical intraepithelial neoplasia: a retrospective, case-control study. Minerva Ginecol. 2017 Oct;69(5):425-430. doi: 10.23736/S0026-4784.17.04053-9. PMID 28675291
- [Background] Chaichian S, Moazzami B, Sadoughi F, Haddad Kashani H, Zaroudi M, Asemi Z. Functional activities of beta-glucans in the prevention or treatment of cervical cancer. J Ovarian Res. 2020 Mar 5;13(1):24. doi: 10.1186/s13048-020-00626-7. PMID 32138756
- [Background] Pietrantoni E, Signore F, Berardi G, Donadio F, Donadio C. [Role of beta-glucan in the treatment of recurrent candidiasis and HPV-correlated lesions and reparative process of epidermis]. Minerva Ginecol. 2010 Feb;62(1):1-5. Italian. PMID 20186110
- [Background] Lavitola G, Della Corte L, De Rosa N, Nappi C, Bifulco G. Effects on Vaginal Microbiota Restoration and Cervical Epithelialization in Positive HPV Patients Undergoing Vaginal Treatment with Carboxy-Methyl-Beta-Glucan. Biomed Res Int. 2020 Apr 27;2020:5476389. doi: 10.1155/2020/5476389. eCollection 2020. PMID 32420349
- [Background] Laccetta G, Carrone A, Burratti M, Mancino P. Effect of the treatment with beta-glucan in women with cervical cytologic report of atypical squamous cells of undetermined significance (ASCUS) and low-grade squamous intraepithelial lesions (L-SIL). Minerva Ginecol. 2015 Apr;67(2):113-20. Epub 2015 Feb 5. PMID 25668505
- [Background] Jentschke M, Lehmann R, Drews N, Hansel A, Schmitz M, Hillemanns P. Psychological distress in cervical cancer screening: results from a German online survey. Arch Gynecol Obstet. 2020 Sep;302(3):699-705. doi: 10.1007/s00404-020-05661-9. Epub 2020 Jun 27. PMID 32594298